CLINICAL TRIAL: NCT04789551
Title: T Cell Profiling in Patients with Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Lifei Hou, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00037843
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Multiple Sclerosis Stable Conditions: Multiple sclerosis patients presenting for a routine clinic visit.
  Interventions: Other: Blood Sample
- Multiple Sclerosis Acute Flare Up: Multiple sclerosis patients admitted to the hospital with acute symptoms.
  Interventions: Other: Blood Sample
- Control patients: Patients without any immunological diseases who present for elective surgery.
  Interventions: Other: Blood Sample

INTERVENTIONS:
Other: Blood Sample — a blood sample will be collected

SUMMARY:
The goal of this research study is to to learn more about the body's immune response in patients with multiple sclerosis (MS). In MS, the body's immune cells mistakenly attack an important part of the nerves of the brain and spinal cord. The immune cells responsible for attacking the nerves in MS patients is primarily the T cells. A marker was recently discovered that might specifically identify these damaging T cells from all other T cells in the body. Understanding which T cells cause the damage in MS patients and understanding more about these specific T cells may help doctors better understand how MS occurs and could possibly prevent MS in the future.

ELIGIBILITY:
MS Group Inclusion criteria

-diagnosis of multiple sclerosis and present to the neurology clinic for a regular checkup or are admitted to the inpatient floor with acute symptoms.

Exclusion criteria

* Have an active infection
* Take T cell modulating drugs

Control Group Inclusion criteria -scheduled for elective surgery

* without any immunological diseases. Exclusion criteria
* Have an active infection.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Multiple Sclerosis who present to Boston Children's Hospital will be enrolled. A group of healthy control patients who present for elective surgery at Boston Children's Hospital will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
T cell populations | up to one week
  compare T cell populations between patients with Multiple Sclerosis and healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hopsital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No